CLINICAL TRIAL: NCT01619007
Title: Xarelto® for Long-term and Initial Anticoagulation in Venous Thromboembolism (VTE)
Brief Title: Treatment of an Acute Deep Vein Thrombosis (DVT) With Either Rivaroxaban or Current Standard of Care Therapy
Acronym: XALIA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 15915; XA1102 (Other: Company Internal)
Record Dates: First submitted 2012-05-29; First posted 2012-06-14 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Deep Vein Thrombosis; Venous Thrombosis
Keywords: Treatment of Venous Thromboembolism; Thromboembolism; Venous Thromboembolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Thromboembolism; Venous Thromboembolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Thrombosis | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Group 2
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Patients who will be treated for an acute deep vein thrombosis (DVT) with rivaroxaban
  Groups: Group 1
Drug: Standard of care — Patients who will be treated for an acute deep vein thrombosis (DVT) with current standard of care comprising e.g. of initial treatment with low-molecular weight heparin or fondaparinux, followed by oral Vitamin-K antagonist for at least 3 months
  Groups: Group 2

SUMMARY:
Following the findings of the clinical trials in drug development, this global non-interventional cohort field study will investigate rivaroxaban under clinical practice conditions in comparison with current standard of care for patients with acute deep vein thrombosis (DVT).

The main goal is to analyze long-term safety in the use of rivaroxaban in the treatment of acute DVT in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients
* Patients >= 18 years
* Patiebts with diagnosis of acute DVT and who have an indication for anticoagulation therapy for at least 12 weeks, who are willing to participate in this study and are available for follow-up

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In- and outpatients in sites participating in the study
Sampling Method: Probability Sample
Enrollment: 5145 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Major bleedings defined as overt bleeding associated with: A fall in hemoglobin of ≥2 g/dL; or a transfusion of ≥2 units of packed red blood cells or whole blood; or occurrence at a critical site | after approximately 2 years or 30 days after stop of therapy
Number of patients with symptomatic recurrent venous thromboembolic events | after approximately 2 years or 30 days after stop of therapy
All cause mortality | after approximately 2 years or 30 days after stop of therapy

SECONDARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse cardiac events collection | after approximately 2 years or 30 days after stop of therapy
Number of patients with other symptomatic thromboembolic events | after approximately 2 years or 30 days after stop of therapy
Treatment satisfaction (patient reported outcomes) | after approximately 2 years or 30 days after stop of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- Many Locations, Austria
- Many Locations, Belgium
- Many Locations, Canada
- Many Locations, Czechia
- Many Locations, Denmark
- Many Locations, France
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Hungary
- Many Locations, Israel
- Many Locations, Italy
- Many Locations, Moldova
- Many Locations, Netherlands
- Many Locations, Norway
- Many Locations, Portugal
- Many Locations, Slovenia
- Many Locations, Spain
- Many Locations, Sweden
- Many Locations, Switzerland
- Many Locations, Ukraine
- Many Locations, United Kingdom

REFERENCES:
- [Derived] Ageno W, Mantovani LG, Haas S, Kreutz R, Monje D, Schneider J, Bugge JP, Gebel M, Turpie AGG. Patient Management Strategies and Long-Term Outcomes in Isolated Distal Deep-Vein Thrombosis versus Proximal Deep-Vein Thrombosis: Findings from XALIA. TH Open. 2019 Mar 26;3(1):e85-e93. doi: 10.1055/s-0039-1683968. eCollection 2019 Jan. PMID 31249987
- [Derived] Ageno W, Mantovani LG, Haas S, Kreutz R, Monje D, Schneider J, van Eickels M, Gebel M, Zell E, Turpie AG. Safety and effectiveness of oral rivaroxaban versus standard anticoagulation for the treatment of symptomatic deep-vein thrombosis (XALIA): an international, prospective, non-interventional study. Lancet Haematol. 2016 Jan;3(1):e12-21. doi: 10.1016/S2352-3026(15)00257-4. Epub 2015 Dec 8. PMID 26765643